CLINICAL TRIAL: NCT03015038
Title: Etude de la réponse Immunitaire Dans l'adénocarcinome Colique
Brief Title: Study of the Immune Response in Colon Adenocarcinoma
Acronym: IMCO
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: C16-21; 2016-A01102-49 (Other: IDRCB)
Record Dates: First submitted 2016-12-12; First posted 2017-01-09 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Colon Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissu and blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Duration of each part of the study per patient:

* Screening: From 1 to 4 weeks
* Sampling period (blood and tissue): 1 day
* Follow-up by patient: 60 months
* Total study duration by patient: 84 months
* Total inclusion duration: 24 months
* Total Follow-up duration: 60 months
* Total study duration: 84 months

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or more.
2. Affiliation to a social security scheme
3. Diagnosis of a colon adenocarcinoma.
4. Patient have signed and dated consent of the study before undertaking procedures related to the study.

Exclusion Criteria:

1. Patients under guardianship / curatorship
2. Following Situations

   * Persons unable to understand, read and / or sign an informed consent
   * Patient with the following functions: investigator or co-investigator, research assistant, pharmacist, study coordinator or having any involvement in the study
   * Uncooperative person or potentially non-compliant for the study and its procedures with predictable difficulties regular monitoring of over 1 year.
   * No affiliation to a social security scheme, a universal medical coverage or any similar plan.
3. Pregnant or lactating women.
4. Patients with HIV seropositivity.
5. Rectal tumor location.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with colon adenocarcinoma treated by surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Immune cells trafficking | Day 0
  Frequency of T cells in the blood and tissue (Flow cytometry method with a panel of Ab).

SECONDARY OUTCOMES:
Infiltration of leucocytes in tumor tissue | Day 0
  Histochemical method with a panel of Ab.
Safety (Number of adverse events, ECOG status) | After Day 0 until the end of the study (Month 3, Month 6, Month 9, Month 12, Month 15, Month 18,Month 21, Month 24, Month 30, Month 36, Month 42, Month 48, Month 54 and Month 60)

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Allez, MD, PhD, Principal Investigator — Hopital Saint Louis
Locations (1):
- Hôpital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonnereau J, Courau T, Asesio N, Salfati D, Bouhidel F, Corte H, Hamoudi S, Hammoudi N, Lavole J, Vivier-Chicoteau J, Chardiny V, Maggiori L, Blery M, Remark R, Bonnafous C, Cattan P, Toubert A, Bhat P, Allez M, Aparicio T, Le Bourhis L. Autologous T cell responses to primary human colorectal cancer spheroids are enhanced by ectonucleotidase inhibition. Gut. 2023 Apr;72(4):699-709. doi: 10.1136/gutjnl-2021-326553. Epub 2022 Jul 8. PMID 35803702
- [Result] Courau T, Bonnereau J, Chicoteau J, Bottois H, Remark R, Assante Miranda L, Toubert A, Blery M, Aparicio T, Allez M, Le Bourhis L. Cocultures of human colorectal tumor spheroids with immune cells reveal the therapeutic potential of MICA/B and NKG2A targeting for cancer treatment. J Immunother Cancer. 2019 Mar 14;7(1):74. doi: 10.1186/s40425-019-0553-9. PMID 30871626